CLINICAL TRIAL: NCT03089619
Title: A Method for Measuring Volume Changes of the Alveolar Ridge During Dental Implantation Using 3D Scanning
Brief Title: Alveolar Management Following Teeth Extraction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties in recruiting of suitable patients, bad compliance of patients
Sponsor: University Medicine Greifswald (Other)
Collaborators: Botiss Medical AG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3D_CHB/collacone; 2015-001434-16 (EudraCT Number)
Record Dates: First submitted 2017-02-27; First posted 2017-03-24 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Alveolar Bone Loss; Bone Resorption
Keywords: Alveolar bone; Bone resorption; dental implants
MeSH Terms: conditions — Alveolar Bone Loss; Bone Resorption

STUDY DESIGN:
Intervention Model Description: assignment of patients to one of the two treatment arms will be carried out randomly. Randomization process will be monitored and carried out by the center of clinical studies coordination - University Medicine Greifswald. Assignment of patient will be only known to the investigator after blood and urine sample results fulfill the inclusion criteria.
Who Masked: Outcomes Assessor
Masking Description: outcome assessors will be masked during the evaluation period. Subjects will be identified through their randomization number. Patients identification log is stored at the study site and only available to the investigator who is responsible of concealment of these information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human-Spongiosa (IMP: drug) (Active Comparator): Product Name: Human-Spongiosa,gefriergetrocknet, CHB / Pharmaceutical form: Granules / Routes of Administration: Dental use / Marketing authorisation number : 3004134.00.00 / Marketing Authorisation Holder: Institute of Transfusion Medicine, Tissue bank, Charité university of medicine Berlin / Used by socket preservation
  Interventions: Drug: Human-Spongiosa
- collacone® (IMP: medical device) (Active Comparator): Product Name: Collacone / Pharmaceutical form: Absorbable, local Hemostat, porcine collagen / Routes of Administration: Dental use / Medical device with a CE mark / Used by socket preservation
  Interventions: Device: collacone®

INTERVENTIONS:
Drug: Human-Spongiosa — after tooth extraction, the dental alveolus is filled with the bone substitute material (Human-Spongiosa) and covered with a membrane (mucoderm®)
  Other Names: Knochenspongiosa of human origin
  Arms: Human-Spongiosa (IMP: drug)
Device: collacone® — after tooth extraction, the dental alveolus is filled with the bone substitute material (collacone®) and covered with a membrane (mucoderm®)
  Other Names: absorbable local hemostat; porcine collagen
  Arms: collacone® (IMP: medical device)

SUMMARY:
Investigation of the volume stability of the alveolar ridge, the bone structure and soft tissue appearance at a delayed dental implantation using two bone substitute materials (1. Human-Spongiosa, gefriergetrocknet, CHB; 2. collacone®)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Indication for tooth extraction resulting in a edentulous gap
* Male and female patients with an age range 20-60 years
* Caucasian
* For female patients: a negative pregnancy test
* Normotonic blood pressure (according to the WHO definition):

  * Men: 110/70 - 140/90 mm Hg
  * Women: 100/60- 140/90mm Hg

Exclusion Criteria:

* Parallel implantation of another implant
* Parallel planned prosthetic restoration of the adjacent teeth
* Smoker (less than 5 years non-smoker)
* Nursing women
* Participation in another clinical trial which dates back to less than 3 months before inclusion in this clinical trial
* Intake of bisphosphonates
* Radiation therapy (medical history or current)
* Known Diabetes mellitus
* Inflammatory processes in the mouth (PSI> 2)
* Presence of autoimmune diseases (Rheumatoid arthritis, Sjögren's syndrome, Systemic lupus erythematosus)
* Presence of blood coagulation disorders (Haemophilia A/B), or the intake of anticoagulants (Warfarin, new oral anticoagulants, aspirin> 100 mg)
* Osteogenesis imperfecta
* Osteoporosis
* Leukemia
* Agranulocytosis
* Immunocompromised patients
* Acute phase and rehabilitation phase of myocardial infarction
* Oncogenes diseases
* Patients undergoing chemotherapy
* Sepsis
* Acute and chronic infections: sinusitis, rhinitis, pharyngitis and Otitis media
* Wound healing disorders
* Seizures
* Gingival hyperplasia
* Alcohol abuse
* Drug abuse
* Infectious diseases (HIV, Hepatitis B and C)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Extent of bone resorption | According to E9 guideline, the assumptions of the sample size calculation and the statistical analysis plan, which was approved by PEI we include "all relevant time points", respective: T-1 (baseline), T2, T3, T5, T6, T7, T8 (see definition above)
  The main objective is to measure the extent of resorption of the alveolar ridge bone following teeth extraction and alveolar management (socket preservation) and to compare the two authorized bone substitute materials:
  1. Human Spongiosa, gefriergetrocknet, CHB + mucoderm® and
  2. collacone® + mucoderm® through 3D surface scan.
  Definition of time points:
  T-1 = baseline T2 = 1 month after extraction T3 = 4.5 months after extraction = time point of implantation T5 = 1 month after implantation T6 = 3 months after implantation T7 = 6 months after implantation T8 = 9 months after implantation

SECONDARY OUTCOMES:
Implants stability | 4.5 months after teeth extraction and socket preservation (T3) and 3 months after implantation (T6)
  The implant stability will be measured 2 times throughout this clinical trial
Pink Esthetic Score | T-1 (baseline before teeth extraction), T1 (7-10 days after extraction), T2 (1 month after extraction), T3 (time of implantation; 4.5 months after extraction), T5, T6, T7 and T8 (respective 1, 3, 6 and 9 months after implantation)
  Repeated measurement of the soft tissues changes throughout the clinical trial at eight times
Histologic bone investigation | 4.5 months after teeth extraction and socket preservation (T3)
  A bone biopsy will be taken before insertion of the implant. The bone biopsy will be investigated for structure changes

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Engeli, Prof., Study Chair — University Greifswald, KKS
Locations (1):
- University Medicine Greifswald - Department for oral and maxillofacial Surgery, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared in accordance with medical data protection regulations.

REFERENCES:
- [Background] Covani U, Ricci M, Bozzolo G, Mangano F, Zini A, Barone A. Analysis of the pattern of the alveolar ridge remodelling following single tooth extraction. Clin Oral Implants Res. 2011 Aug;22(8):820-5. doi: 10.1111/j.1600-0501.2010.02060.x. Epub 2010 Dec 29. PMID 21198897
- [Background] Morjaria KR, Wilson R, Palmer RM. Bone healing after tooth extraction with or without an intervention: a systematic review of randomized controlled trials. Clin Implant Dent Relat Res. 2014 Feb;16(1):1-20. doi: 10.1111/j.1708-8208.2012.00450.x. Epub 2012 Mar 8. PMID 22405099
- [Background] Fiorellini JP, Howell TH, Cochran D, Malmquist J, Lilly LC, Spagnoli D, Toljanic J, Jones A, Nevins M. Randomized study evaluating recombinant human bone morphogenetic protein-2 for extraction socket augmentation. J Periodontol. 2005 Apr;76(4):605-13. doi: 10.1902/jop.2005.76.4.605. PMID 15857102
- [Background] Kernan WN, Viscoli CM, Makuch RW, Brass LM, Horwitz RI. Stratified randomization for clinical trials. J Clin Epidemiol. 1999 Jan;52(1):19-26. doi: 10.1016/s0895-4356(98)00138-3. PMID 9973070
- [Background] Harrell FE, Jr. Regression Modeling Strategies. With Applications to Linear Models, Logistic and Ordinal Regression, and Survival Analysis. 2nd ed. Heidelberg: Springer; 2015
- [Background] Schafer JL, Graham JW. Missing data: our view of the state of the art. Psychol Methods. 2002 Jun;7(2):147-77. PMID 12090408
- [Background] Cardaropoli G, Araujo M, Lindhe J. Dynamics of bone tissue formation in tooth extraction sites. An experimental study in dogs. J Clin Periodontol. 2003 Sep;30(9):809-18. doi: 10.1034/j.1600-051x.2003.00366.x. PMID 12956657
- [Background] Schwarz F, Rothamel D, Ferrari D, Becker J. Aktuelle Aspekte zur Beeinflussung der Dimensionsveränderung des Alveolarknochens nach Zahnentfernung Implantologie 14 Vol 42006:319-333.
- [Background] Amler MH. The time sequence of tissue regeneration in human extraction wounds. Oral Surg Oral Med Oral Pathol. 1969 Mar;27(3):309-18. doi: 10.1016/0030-4220(69)90357-0. No abstract available. PMID 5251474
- [Background] Kuboki Y, Hashimoto F, Ishibashi K. Time-dependent changes of collagen crosslinks in the socket after tooth extraction in rabbits. J Dent Res. 1988 Jun;67(6):944-8. doi: 10.1177/00220345880670061101. PMID 3170907
- [Background] Lin WL, McCulloch CA, Cho MI. Differentiation of periodontal ligament fibroblasts into osteoblasts during socket healing after tooth extraction in the rat. Anat Rec. 1994 Dec;240(4):492-506. doi: 10.1002/ar.1092400407. PMID 7879901
- [Background] Cardaropoli G, Araujo M, Hayacibara R, Sukekava F, Lindhe J. Healing of extraction sockets and surgically produced - augmented and non-augmented - defects in the alveolar ridge. An experimental study in the dog. J Clin Periodontol. 2005 May;32(5):435-40. doi: 10.1111/j.1600-051X.2005.00692.x. PMID 15842256
- [Background] Schropp L, Kostopoulos L, Wenzel A, Isidor F. Clinical and radiographic performance of delayed-immediate single-tooth implant placement associated with peri-implant bone defects. A 2-year prospective, controlled, randomized follow-up report. J Clin Periodontol. 2005 May;32(5):480-7. doi: 10.1111/j.1600-051X.2005.00699.x. PMID 15842263
- [Background] Fickl S, Schneider D, Zuhr O, Hinze M, Ender A, Jung RE, Hurzeler MB. Dimensional changes of the ridge contour after socket preservation and buccal overbuilding: an animal study. J Clin Periodontol. 2009 May;36(5):442-8. doi: 10.1111/j.1600-051X.2009.01381.x. PMID 19419446
- [Background] Lundgren D, Sennerby L, Falk H, Friberg B, Nyman S. The use of a new bioresorbable barrier for guided bone regeneration in connection with implant installation. Case reports. Clin Oral Implants Res. 1994 Sep;5(3):177-84. doi: 10.1034/j.1600-0501.1994.050309.x. PMID 7827233
- [Background] Polson AM, Garrett S, Stoller NH, Greenstein G, Polson AP, Harrold CQ, Laster L. Guided tissue regeneration in human furcation defects after using a biodegradable barrier: a multi-center feasibility study. J Periodontol. 1995 May;66(5):377-85. doi: 10.1902/jop.1995.66.5.377. PMID 7623257
- [Background] Laurell L, Falk H, Fornell J, Johard G, Gottlow J. Clinical use of a bioresorbable matrix barrier in guided tissue regeneration therapy. Case series. J Periodontol. 1994 Oct;65(10):967-75. doi: 10.1902/jop.1994.65.10.967. PMID 7823279
- [Background] Lekovic V, Camargo PM, Klokkevold PR, Weinlaender M, Kenney EB, Dimitrijevic B, Nedic M. Preservation of alveolar bone in extraction sockets using bioabsorbable membranes. J Periodontol. 1998 Sep;69(9):1044-9. doi: 10.1902/jop.1998.69.9.1044. PMID 9776033
- [Background] Shakibiae M. Alveolenmanagement nach Zahnextraktion - Socket und Ridge Preservation. Dental Magazin Vol 22009:24-33.
- [Background] Hammerle CH, Jung RE, Yaman D, Lang NP. Ridge augmentation by applying bioresorbable membranes and deproteinized bovine bone mineral: a report of twelve consecutive cases. Clin Oral Implants Res. 2008 Jan;19(1):19-25. doi: 10.1111/j.1600-0501.2007.01407.x. Epub 2007 Oct 22. PMID 17956571
- [Background] Araujo MG, Lindhe J. Ridge preservation with the use of Bio-Oss collagen: A 6-month study in the dog. Clin Oral Implants Res. 2009 May;20(5):433-40. doi: 10.1111/j.1600-0501.2009.01705.x. PMID 19522974
- [Background] Mardas N, Chadha V, Donos N. Alveolar ridge preservation with guided bone regeneration and a synthetic bone substitute or a bovine-derived xenograft: a randomized, controlled clinical trial. Clin Oral Implants Res. 2010 Jul;21(7):688-98. doi: 10.1111/j.1600-0501.2010.01918.x. PMID 20636724
- [Background] Nevins M, Camelo M, De Paoli S, Friedland B, Schenk RK, Parma-Benfenati S, Simion M, Tinti C, Wagenberg B. A study of the fate of the buccal wall of extraction sockets of teeth with prominent roots. Int J Periodontics Restorative Dent. 2006 Feb;26(1):19-29. PMID 16515093
- [Background] Friedman LM, Furberg CD, DeMets DL, Reboussin DM, Granger CB. Fundamentals of Clinical Trials. 5th ed. Heidelberg: Springer; 2015.
- [Background] Greenland S, Poole C. Living with p values: resurrecting a Bayesian perspective on frequentist statistics. Epidemiology. 2013 Jan;24(1):62-8. doi: 10.1097/EDE.0b013e3182785741. PMID 23232611
- [Background] Enkling N, Bayer S, Johren P, Mericske-Stern R. Vinylsiloxanether: a new impression material. Clinical study of implant impressions with vinylsiloxanether versus polyether materials. Clin Implant Dent Relat Res. 2012 Mar;14(1):144-51. doi: 10.1111/j.1708-8208.2009.00240.x. Epub 2009 Sep 29. PMID 19793332
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Feng SW, Chang WJ, Lin CT, Lee SY, Teng NC, Huang HM. Modal damping factor detected with an impulse-forced vibration method provides additional information on osseointegration during dental implant healing. Int J Oral Maxillofac Implants. 2015 Nov-Dec;30(6):1333-40. doi: 10.11607/jomi.4038. PMID 26574858
- [Background] Witte F, Ulrich H, Palm C, Willbold E. Biodegradable magnesium scaffolds: Part II: peri-implant bone remodeling. J Biomed Mater Res A. 2007 Jun 1;81(3):757-65. doi: 10.1002/jbm.a.31293. PMID 17390322